CLINICAL TRIAL: NCT01502956
Title: Refractory Overactive Bladder: Sacral NEuromodulation v. BoTulinum Toxin Assessment (ROSETTA)
Acronym: ROSETTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: Duke University (Other); University of Alabama at Birmingham (Other); University of California, San Diego (Other); The Cleveland Clinic (Other); Brown University (Other); University of New Mexico (Other); University of Pennsylvania (Other); University of Pittsburgh (Other); Oregon Health and Science University (Other); RTI International (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PFDN 20; U01HD069031 (NIH)
Record Dates: First submitted 2011-12-27; First posted 2012-01-02 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Urinary Incontinence, Urge
Keywords: Refractory Urinary Urge Incontinence; Botox A®; Interstim® Device
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- InterStim® device (Active Comparator): The FSLP InterStim® device is to be done within 3 months of enrolling/consenting. The 1st stage is lead placement into the S3 foramen with best response to stimulation. The 4 electrodes will be tested and set to an amplitude that achieves comfortable stimulation in the vaginal, perineal, or rectal sensation. If =/>50% improvement, participant will then have the 2nd stage IPG implantation, 8-18 days after last FSLP. If there is a technical problem with lead on 1st FSLP, then the participant can have a 2nd FSLP and may go on to have IPG implantation with lead replacement. The 2nd FSLP must be initiated no longer than 1 month since the initiation of the 1st FSLP. If the participant is a non-responder and there is no technical problem, then the lead is removed.
  Interventions: Device: InterStim® device
- Botox® injection (Active Comparator): Total of 200 units of Botox A will be dissolved into 10mL of saline and injected into the bladder within 3 months of enrolling/consenting. Participants determined to have a clinical response at the 1 month visit (post 1st injection) may receive additional injections between 6-24 months.
  Interventions: Drug: Botox® injection

INTERVENTIONS:
Device: InterStim® device — Eligible subjects will complete baseline assessments, be randomized and scheduled for first stage lead placement (FSLP) InterStim®. The criterion for an initial clinical response to InterStim® therapy will be defined as a ≥50% improvement in the mean number of UUIE/day on a minimum 3 day bladder diary, completed during the 7-14 days following the first stage lead placement (FSLP). Subjects with a ≥ 50% improvement mean number of UUIE/day will be eligible to proceed with implantation of the implantable pulse generator (IPG). Subjects will then be followed monthly to determine the response to therapy.
  Arms: InterStim® device
Drug: Botox® injection — Eligible subjects will complete baseline assessments, be randomized and scheduled for Botox A® injection visit. Subjects who received a Botox A® injection will be assessed for a clinical response, at 1 month from injection, using the same clinical criterion (≥50% improvement in the mean number of UUIE/day on a 3 day bladder diary completed prior to the 1 month visit). Those subjects that experience a clinical response, at one month, will be eligible for a repeat Botox A® injection after 6 months, if they experience degradation of clinical effect, using the PGSC.
  Other Names: Botox
  Arms: Botox® injection

SUMMARY:
The purpose of this randomized, open-label, active-control trial is to compare the effectiveness of intra-detrusor botulinum toxin A (Botox A®, Allergan) versus sacral neuromodulation (InterStim®, Medtronic) for the treatment of refractory urge urinary incontinence. In addition, the study will evaluate select technical attributes of the interventions as well as the effect of these two interventions on other lower urinary tract and pelvic floor symptoms.

Hypothesis: InterStim® therapy will result in a greater reduction in daily urge urinary incontinence episodes over the 6-month follow-up period as compared to Botox A® injection.

A supplemental study investigates whether biological markers including those related to inflammation and connective tissue remodeling change following treatments with Botox A® and Interstim®.

DETAILED DESCRIPTION:
Primary Aim:

To compare the change from baseline in the number of urge urinary incontinence episodes (UUIE) over 6 the six month follow-up period in women randomized to sacral neuromodulation (InterStim®) therapy, versus those randomized to intra-detrusor injection with 200 units of botulinum toxin A (Botox A®).

Secondary Aims:

* Long Term Efficacy: To compare the long-term (12 and 24 month) efficacy outcomes in women randomized to sacral neuromodulation(InterStim®) therapy, versus those randomized to intra-detrusor injection with 200 units of botulinum toxin A (Botox A®). Secondary efficacy outcomes, collected at 12 and 24 months as well as 6 months,include adequate control of their urge urinary incontinence, change in bothersome symptoms of urinary urge incontinence (UUI), severity of urge incontinence, urinary frequency, nocturia, subject satisfaction with therapy, quality of life measures and bowel and sexual function.
* Cost Effectiveness: To compare utilization of medical resources for cost effectiveness analysis and cost-utility between treatment groups.
* Treatment Safety and Burden: To assess safety profile and treatment burden of both interventions by comparing adverse event incidence between treatment arms, and also by obtaining estimates of incidence of treatment-specific safety and burden outcomes. Safety and burden outcomes for Botox A® injections include receipt of additional injections and intermittent catheterization due to voiding dysfunction/partial urinary retention. Safety and burden outcomes for InterStim® device include infection, pain, lead migration, reprogramming (and reasons for) and surgical revision (and reasons for).

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adult female at least 21 years old, with no plans to become pregnant during the course of the trial) and if of child-bearing potential, with a negative pregnancy test, and if sexually active, must be using medically acceptable contraception.
* 6 urge urinary incontinence episodes on a 3-day baseline bladder diary, with these urge incontinence episodes representing greater than 50% of the total incontinent episodes recorded.
* Willing and able to complete all study related items and interviews.
* Refractory urinary urge urinary incontinence: defined as (1) Persistent symptoms despite at least one or more conservative treatments (e.g. supervised behavioral therapy, supervised physical therapy); and (2)Persistent symptoms despite the use of a minimum of two anticholinergics, or unable to tolerate medication due to side effects, or has a contraindication to taking anticholinergic medication.
* Currently not on an anticholinergic or antimuscarinic medication (e.g. oxybutynin, tolterodine, and/or fesoterodine) or be willing to stop medication for 3 weeks prior to completing baseline bladder diary and expected to remain off medications through duration of study.
* Demonstrates ability (or have caregiver demonstrate ability) to perform clean intermittent self-catheterization.
* Grossly neurologically normal on exam and no gross systemic neurologic conditions believed to affect urinary function.
* Urodynamic assessment within the previous 18 months prior to enrollment or done after enrollment, prior to randomization.

Exclusion Criteria:

* Neurologic diseases such as multiple sclerosis, Parkinson Disease, CVA within 6 months prior to enrollment, myasthenia gravis, Charcot-Marie-Tooth disease, clinically significant peripheral neuropathy, and complete spinal cord injury.
* Untreated urinary tract infection (UTI).
* Any prior use of either study therapy for treatment of urinary urge incontinence (Botox A® or Interstim®).
* Current participation in any other conflicting interventional research study.
* PVR >150 ml on 2 occasions within 6 months prior to enrollment (If the PVR value was obtained by ultrasound and was ≥150 ml, the PVR will be confirmed by catheterization which will be the gold standard)
* Subjects with knowledge of planned MRIs or diathermy, except those allowable per Medtronic guidelines.
* Current or prior bladder malignancy.
* Surgically altered detrusor muscle, such as augmentation cystoplasty.
* Subjects taking aminoglycosides.
* Currently pregnant or lactating.
* Subjects who are on ambulatory anticoagulant therapy, including aspirin, who are unable to discontinue treatment for 24 hours prior to bladder injection and staged InterStim® procedure.
* Serum creatinine level greater than twice the upper limit of normal within the previous year prior to enrollment.
* Surgical treatment for stress incontinence (sling, Burch or urethral injection) or pelvic organ prolapse recommended or planned at enrollment by study investigator(s).
* Prior stress incontinence or prolapsed surgery within the last 6 months prior to enrollment.
* Allergy to lidocaine or bupivacaine.
* Prior pelvic radiation.
* Uninvestigated hematuria.
* Greater than or equal to Stage III vaginal prolapse.
* Known allergy to Botox A®.
* Use of a vaginal pessary.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2012-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Amundsen, MD, Study Chair — Duke University; Holly Richter, PhD, MD, Principal Investigator — University of Alabama at Birmingham; Shawn A. Menefee, MD, Principal Investigator — Kaiser Permanente, San Diego, CA; Sandip Vasada, MD, Principal Investigator — The Cleveland Clinic; Deborah L. Myers, MD, Principal Investigator — Brown/Women and Infants Hospital of Rhode Island; Yoko Kumesu, MD, Principal Investigator — University of New Mexico; Lily Arya, MD, Principal Investigator — University of Pennsylvania; Jerry Lowder, MD, Principal Investigator — University of Pittsburgh; W. Thomas Gregory, MD, Principal Investigator — Oregon Health and Science University; Dennis Wallace, PhD, Principal Investigator — RTI International; Susan Meikle, MD, MSPH, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Department of Obstetrics and Gynecology, Birmingham, Alabama
  - University of California, San Diego, Women's Pelvic Medicine Center, La Jolla, California
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Duke Division of Urogynecology and Reconstructive Pelvic Surgery, Durham, North Carolina
  - Cleveland Clinic, Obstretric and Gynecology and Women Health Institute, Cleveland, Ohio
  - Oregon Health and Science University, Kohler Pavilion, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Univesity of Pittsburgh, Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Center for Women's Pelvic Medicine and Reconstructive Surgery, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hendrickson WK, Amundsen CL, Rahn DD, Meyer I, Bradley MS, Smith AL, Myers DL, Jelovsek JE, Lukacz ES. Comparison of 100 U With 200 U of Intradetrusor OnabotulinumToxinA for Nonneurogenic Urgency Incontinence. Female Pelvic Med Reconstr Surg. 2021 Mar 1;27(3):140-146. doi: 10.1097/SPV.0000000000001020. PMID 33620895
- [Derived] Richter HE, Jelovsek JE, Iyer P, Rogers RG, Meyer I, Newman DK, Bradley MS, Harm-Ernandes I, Dyer KY, Wohlrab K, Mazloomdoost D, Gantz MG; Eunice Kennedy Shriver NICHD Pelvic Floor Disorders Network and the National Institutes of Health Office of Research on Women's Health. Characteristics Associated With Clinically Important Treatment Responses in Women Undergoing Nonsurgical Therapy for Fecal Incontinence. Am J Gastroenterol. 2020 Jan;115(1):115-127. doi: 10.14309/ajg.0000000000000482. PMID 31895722
- [Derived] Andy UU, Amundsen CL, Honeycutt E, Markland AD, Dunivan G, Dyer KY, Korbly NB, Bradley M, Vasavada S, Mazloomdoost D, Thomas S; NICHD Pelvic Floor Disorders Network. Sacral neuromodulation versus onabotulinumtoxinA for refractory urgency urinary incontinence: impact on fecal incontinence symptoms and sexual function. Am J Obstet Gynecol. 2019 Nov;221(5):513.e1-513.e15. doi: 10.1016/j.ajog.2019.06.018. Epub 2019 Jun 15. PMID 31211964
- [Derived] Komesu YM, Amundsen CL, Richter HE, Erickson SW, Ackenbom MF, Andy UU, Sung VW, Albo M, Gregory WT, Paraiso MF, Wallace D; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network. Refractory urgency urinary incontinence treatment in women: impact of age on outcomes and complications. Am J Obstet Gynecol. 2018 Jan;218(1):111.e1-111.e9. doi: 10.1016/j.ajog.2017.10.006. Epub 2017 Oct 12. PMID 29031894
- [Derived] Amundsen CL, Richter HE, Menefee S, Vasavada S, Rahn DD, Kenton K, Harvie HS, Wallace D, Meikle S. The Refractory Overactive Bladder: Sacral NEuromodulation vs. BoTulinum Toxin Assessment: ROSETTA trial. Contemp Clin Trials. 2014 Mar;37(2):272-83. doi: 10.1016/j.cct.2014.01.009. Epub 2014 Jan 30. PMID 24486637

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women who have persistent severe UUI symptoms, defined as ≥6 UUI episodes on a 3-day bladder diary are recruited from urology and urogynecology subspecialty clinics as well as by other marketing methods.
Groups:
- InterStim® Device: The FSLP InterStim® device is to be done within 3 months of enrolling/consenting. The 1st stage is lead placement into the S3 foramen with best response to stimulation. The 4 electrodes will be tested and set to an amplitude that achieves comfortable stimulation in the vaginal, perineal, or rectal sensation. If =/>50% improvement, participant will then have the 2nd stage IPG implantation, 8-18 days after last FSLP. If there is a technical problem with lead on 1st FSLP, then the participant can have a 2nd FSLP and may go on to have IPG implantation with lead replacement. The 2nd FSLP must be initiated no longer than 1 month since the initiation of the 1st FSLP. If the participant is a non-responder and there is no technical problem, then the lead is removed.
  InterStim® device: Eligible subjects will complete baseline assessments, be randomized and scheduled for first stage lead placement (FSLP) InterStim®. The criterion for an initial clinical response to InterStim® therapy will be d
Period: Overall Study
Arm/Group | InterStim® Device | Botox® Injection
Started | 192 | 194
Completed | 168 | 168
Not Completed | 24 | 26
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 14 | 11
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 8 | 10

BASELINE CHARACTERISTICS:
Population: All eligible participants who provided at least 1 post-baseline diary assessment.
Groups:
- InterStim® Device: The FSLP InterStim® device is to be done within 3 months of enrolling/consenting. The 1st stage is lead placement into the S3 foramen with best response to stimulation. The 1st stage is lead placement into the S3 foramen with best response to stimulation.The 4 electrodes will be tested and set to an amplitude that achieves comfortable stimulation in the vaginal, perineal, or rectal sensation. If =/>50% improvement, participant will then have the 2nd stage IPG implantation, 8-18 days after last FSLP. If there is a technical problem with lead on 1st FSLP, then the participant can have a 2nd FSLP and may go on to have IPG implantation with lead replacement. The 2nd FSLP must be initiated no longer than 1 month since the initiation of the 1st FSLP. If the participant is a non-responder and there is no technical problem, then the lead is removed.
- Total: Total of all reporting groups
Arm/Group | InterStim® Device | Botox® Injection | Total
Number analyzed (Participants) | 174 | 190 | 364
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (11.8) | 62.9 (11.5) | 63.0 (11.6)
Age, Customized [Count of Participants; unit: Participants]
  Age <65 years | 91 | 100 | 191
  Age => 65 years | 83 | 90 | 173
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 174 | 190 | 364
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 18 | 28
  Not Hispanic or Latino | 160 | 167 | 327
  Unknown or Not Reported | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 149 | 154 | 303
  Black | 16 | 22 | 38
  American Indian/Alaska Native | 1 | 4 | 5
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 7 | 9 | 16
Menopausal Status [Count of Participants; unit: Participants]
  Pre-menopausal | 18 | 20 | 38
  Post-menopausal | 149 | 162 | 311
  Not sure | 7 | 8 | 15
History of Recurrent UTIs [Count of Participants; unit: Participants]
  No history of recurrent UTIs | 149 | 166 | 315
  History of recurrent UTIs | 25 | 24 | 49
Urinary Incontinence Episodes Per Day [Mean (Standard Deviation); unit: Episodes per day]
  Total incontinence episodes per day | 5.8 (3.0) | 6.0 (3.0) | 5.9 (3.0)
  Urge incontinence episodes per day | 5.2 (2.7) | 5.4 (2.7) | 5.3 (2.7)
Nocturia (number of night voids per day) [Mean (Standard Deviation); unit: Voids per day] | 1.7 (1.4) | 1.7 (1.2) | 1.7 (1.3)
Overactive Bladder Questionnaire - Short Form (OABq-SF) [Mean (Standard Deviation); unit: units on a scale] — Values range from 0 to 100 with higher scores on the symptom scale indicating greater severity of symptoms and higher scores on the quality of life scale indicating better quality of life.
  units on a scale
    OABq-SF Symptom Bother | 76.1 (16.8) | 74.6 (19.5) | 75.3 (18.3)
    OABq-SF Quality of Life | 36.8 (21.6) | 38.2 (23.0) | 37.5 (22.3)
Urinary Frequency and Nocturia - Sandvik Questionnaire [Count of Participants; unit: Participants] — Patient-reported measure of incontinence severity as assessed on a scale of slight (1-2) to very severe (10-12) using the standard scoring algorithm.
  Participants
    Slight | 1 | 2 | 3
    Moderate | 25 | 27 | 52
    Severe | 38 | 52 | 90
    Very Severe | 105 | 103 | 208
Urinary Distress Inventory Short Form (UDI-SF) [Mean (Standard Deviation); unit: units on a scale] — Values range from 0 to 100 with higher scores indicating greater distress.
  units on a scale | 59.2 (16.9) | 60.9 (18.3) | 60.1 (17.7)
Incontinence Impact Questionnaire Short Form (IIQ-SF) [Mean (Standard Deviation); unit: units on a scale] — Values range from 0 to 100 with higher scores indicating worse quality of life.
  units on a scale | 52.5 (25.8) | 52.7 (27.6) | 52.6 (26.7)
Health Utilities Index Mark 3 (HUI-3) [Mean (Standard Deviation); unit: units on a scale] — Values are defined such that the score for dead is 0; the score for perfect health is 1.0.
  units on a scale | 0.74 (0.28) | 0.71 (0.30) | 0.73 (0.29)

OUTCOME MEASURES:

1. Primary Outcome: Number of Urge Urinary Incontinence (UUI) Episodes
Description: The primary outcome is the change from baseline in mean number of UUI episodes over the first 6-month visit period (1, 2, 3, 4, 5 and 6 month assessments); and is measured using 3-day bladder diaries administered monthly for the first 6 month visit period.
Time Frame: 6 Months
Population: All eligible participants who provided at least 1 post-baseline diary assessment.
Measure: Mean (95% Confidence Interval); unit: UUI episodes
Arm/Group | InterStim® Device | Botox® Injection
Number analyzed (Participants) | 174 | 190
UUI episodes | -3.25 [-3.64 to -2.87] | -3.89 [-4.26 to -3.52]

2. Secondary Outcome: Number of Participants With Improvement of Bladder Function and Urinary Leakage
Description: Proportion of subjects who report adequate improvement of their bladder function and urinary leakage with the Patient Global Impression of Improvement Questionnaire (PGI-I) at 6 months. Adequate improvement is defined as a rating of 1, 2, or 3 (better) on the patient-reported measure of perceived improvement with treatment on a scale of 1 (very much better) to 7 (very much worse).
Time Frame: 6 Months
Population: All eligible participants who provided at least 1 postbaseline diary assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | InterStim® Device | Botox® Injection
Number analyzed (Participants) | 174 | 190
Participants
  Urinary leakage | 91 | 101
  Bladder function | 92 | 100

3. Secondary Outcome: Change in Overactive Bladder
Description: Change in mean Overactive Bladder Questionnaire Short Form (OABq-SF) score throughout baseline to the first 6-month visit (1, 2, 3, 4, 5, and 6-month assessments). Values range from 0 to 100 with higher scores on the symptom scale indicating greater severity of symptoms and higher scores on the quality of life scale indicating a better quality of life.
Time Frame: 6 Months
Population: All eligible participants who provided at least 1 post-baseline diary assessment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | InterStim® Device | Botox® Injection
Number analyzed (Participants) | 174 | 190
units on a scale
  OABq-SF Symptom Bother | -38.6 [-42.5 to -34.6] | -46.7 [-50.5 to -43.0]
  OABq-SF Quality of Life | 38.1 [34.1 to 42.0] | 41.6 [37.9 to 45.4]

4. Secondary Outcome: Urinary Frequency and Nocturia
Description: Change in mean number of urinary incontinence episodes (any type) and nocturia episodes from baseline over the first 6-month visit period (1, 2, 3, 4, 5, and 6-month assessments) as measured by the 3 day bladder diary.
Time Frame: 6 Months
Population: All eligible participants who provided at least 1 post-baseline diary assessment.
Measure: Mean (95% Confidence Interval); unit: Number of episodes
Arm/Group | InterStim® Device | Botox® Injection
Number analyzed (Participants) | 174 | 190
Number of episodes
  Incontinence episodes (any) | -3.50 [-3.94 to -3.06] | -4.02 [-4.44 to -3.61]
  Nocturia episodes | -0.26 [-0.43 to -0.10] | -0.40 [-0.56 to -0.24]

5. Secondary Outcome: Severity of Urge Incontinence Symptoms
Description: Severity of urge incontinence symptoms at 6 month visit period as measured by the Sandvik questionnaire. The Sandvik score is a patient-reported measure of incontinence severity as assessed on a scale of slight (1-2), moderate (3-6), severe (8-9), very severe (12) to severe (10-12) using a standard scoring algorithm.
Time Frame: 6 Months
Population: All eligible participants who provided at least 1 post-baseline diary assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | InterStim® Device | Botox® Injection
Number analyzed (Participants) | 174 | 190
Participants
  Sandvik Slight | 23 | 29
  Sandvik Moderate | 33 | 33
  Sandvik Severe | 24 | 28
  Sandvik Very Severe | 44 | 36

6. Secondary Outcome: Treatment Satisfaction (OAB-SATq Treatment Satisfaction, Adverse Effects, Treatment Endorsement, and Convenience)
Description: Treatment satisfaction as measured by the mean Overactive Bladder Satisfaction of Treatment Questionnaire (OAB-SATq) score at 6 months (6 month assessment). The OAB-SATq score ranges from 0 to 100 and includes 5 subscales: treatment satisfaction, side effects, treatment endorsement, convenience, and treatment preference, with higher scores reflecting better satisfaction.
Time Frame: 6 months
Population: All eligible participants who provided at least 1 post-baseline diary assessment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | InterStim® Device | Botox® Injection
Number analyzed (Participants) | 174 | 190
units on a scale
  OAB-SATq Treatment Satisfaction | 59.8 [55.0 to 64.7] | 67.7 [63.2 to 72.1]
  OAB-SATq Adverse Effects | 85.1 [81.1 to 89.2] | 88.4 [84.7 to 92.2]
  OAB-SATq Endorsement | 67.6 [62.9 to 72.3] | 78.1 [73.7 to 82.4]
  OAB-SATq Convenience | 70.2 [65.8 to 74.5] | 67.6 [63.7 to 71.6]

7. Secondary Outcome: Treatment Satisfaction (OAB-SATq Treatment Preference)
Description: Treatment preference as measured by the Overactive Bladder Satisfaction of Treatment Questionnaire (OAB-SATq) at 6 months (6 month assessment).OAB-SATq treatment preference is a binary outcome that is classified as yes if a participant answers either "Slight preference for the treatment I am receiving now" or "Definitely prefer the treatment I am receiving now" to the question "Do you prefer the treatment that you received since entering this study to the treatment you received before the study?"
Time Frame: 6 Months
Population: All eligible participants who provided at least 1 postbaseline diary assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | InterStim® Device | Botox® Injection
Number analyzed (Participants) | 174 | 190
Participants | 89 | 113

8. Secondary Outcome: Quality of Life (UDI-SF)
Description: Change from baseline in quality of life measures over the first 6 month visit period (6 month assessment) as measured by the change in mean Urinary Distress Inventory Short Form (UDI-SF) score. The UDI-SF scale has a range from 0 to 100 with higher scores indicating greater distress.
Time Frame: 6 Months
Population: All eligible participants who provided at least 1 post-baseline diary assessment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | InterStim® Device | Botox® Injection
Number analyzed (Participants) | 174 | 190
units on a scale | -8.6 [-10.9 to -6.3] | -10.0 [-12.2 to -7.8]

9. Secondary Outcome: Quality of Life (IIQ-SF)
Description: Change from baseline in quality of life measures over the first 6 month visit period (6 month assessment) as measured by the change in the mean Incontinence Impact Questionnaire short form (IIQ-SF) score. The IIQ-SF scale has a range from 0 to 100 with higher scores indicating a worse quality of life.
Time Frame: 6 Months
Population: All eligible participants who provided at least 1 post-baseline diary assessment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | InterStim® Device | Botox® Injection
Number analyzed (Participants) | 174 | 190
units on a scale | -10.4 [-13.0 to -7.8] | -12.4 [-14.9 to -9.9]

10. Secondary Outcome: Quality of Life (HUI-3)
Description: Change from baseline in quality of life measures over the first 6 month visit period (6 month assessment) as measured by the Health Utility Index, Version 3 (HUI-3). The HUI 3 scale has a range from 0 to 1 with higher scores representing better health.
Time Frame: 6 Months
Population: All eligible participants who provided at least 1 post-baseline diary assessment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | InterStim® Device | Botox® Injection
Number analyzed (Participants) | 174 | 190
units on a scale | -0.006 [-0.025 to 0.013] | -0.011 [-0.028 to 0.007]

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting on or after day 0 and on or before 6-month visit.
Description: If a subject experienced more than 1 of a given AE, the subject is counted only once for that AE.
Arm/Group | InterStim® Device | Botox® Injection
Serious Adverse Events (participants affected / at risk) | 58/178 | 58/191
Other Adverse Events (participants affected / at risk) | 20/178 | 66/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | InterStim® Device (N=178) | Botox® Injection (N=191)
Abscess (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 2 (4) | 0 (0)
Clostridium difficile sepsis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 4 (4)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (2)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Abdominal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Anal sphincterotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Endotracheal intubation (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Hernia hiatus repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Intestinal resection (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 2 (2)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Mammoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device change (Surgical and medical procedures) | 2 (2) | 0 (0)
Medical device removal (Surgical and medical procedures) | 3 (3) | 0 (0)
Skin graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Tenotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (5) | 2 (3)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 2 (2)
Device deployment issue (General disorders) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 3 (3) | 0 (0)
Hernia (General disorders) | 1 (1) | 1 (1)
Medical device site pain (General disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cyst aspiration (Investigations) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Sexual abuse (Social circumstances) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | InterStim® Device (N=178) | Botox® Injection (N=191)
Urinary Tract Infection (Infections and infestations) | 20 (28) | 66 (107)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No